CLINICAL TRIAL: NCT01229202
Title: Use of Vascular Endothelial Growth Factor Inhibitor, Bevacizumab to Modulate the Outcomes of Trabeculectomy Surgery
Brief Title: Use of Bevacizumab to Modulate the Outcomes of Trabeculectomy Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No REB file
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CD-2007-331
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2022-10

CONDITIONS: Glaucoma
Keywords: trabeculectomy; glaucoma surgery; bevacizumab; Vascular Endothelial Growth Inhibitor; glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard of care (Active Comparator): standard of care for trabeculectomy surgery
  Interventions: Drug: Bevacizumab
- bevacizumab arm (Active Comparator)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — single bevacizumab subtenon injection of 1.25 mg. at end of trabeculectomy surgery
  Other Names: Avastin

SUMMARY:
Vascular epithelial growth factor (VEGF) plays a critical role in vessel growth and wound healing. Bevacizumab, a non specific VEGF inhibitor, has been successfully used for the treatment of eye diseases associated with neovascularization. The purpose of this randomized study is 1) to investigate the effects of intraoperative subtenon injection of bevacizumab on the outcomes of trabeculectomy surgery. 2) to measure plasma and aqueous levels of VEGF and assess its association with the outcomes of trabeculectomy surgery. Trabeculectomy surgery, where a small drainage canal is created at the front of the eye, is the most common glaucoma surgery performed worldwide. The goal of the surgery is to control intraocular pressure. Failure of this procedure is most commonly caused by excessive scarring of the surgical site. If scarring occurs, the drainage canal can close. By adding Bevacizumab at the time of surgery, wound healing may be slowed and surgical failure prevented.

The results of this study will be helpful in the future development of new more effective and safe surgical techniques for treatment of glaucoma.

Patients who have given informed consent are randomized into two groups. One group receives standard of care for trabeculectomy surgery and the other group receives standard of care plus an injection of Bevacizumab at the surgery site. Both groups have a one time collection of ocular fluid and a blood sample taken from a vein in the arm. After surgery, patients are seen by their study doctor six times in the following year. At these visits measurements are taken of their visual acuity, eye pressure and blood pressure. The doctor does a clinical exam and at months six and twelve photographs of the patients' eye are taken.

ELIGIBILITY:
Inclusion Criteria:

* any type of glaucoma, except neovascular or inflammatory
* patients requiring trabeculectomy or combined cataract surgery with trabeculectomy surgery

Exclusion Criteria:

* younger than 30 years of age
* previous ocular surgeries excepting cataract surgeries
* patients who have had or present with intraocular inflammation
* neovascular glaucoma
* patients who are aphakic
* diabetic retinopathy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07 (Estimated); Primary Completion 2012-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
post surgery IOP (Intra Ocular Pressure Measurement) | one year post surgery

SECONDARY OUTCOMES:
bleb appearance | one year post surgery
number of bleb needlings | one year post surgery
number of glaucoma medications at 12 months postoperatively | one year post surgery
eye complications | one year post surgery
systemic complications | one year post surgery
need for another glaucoma surgery to control glaucoma | one year post surgery
postoperative visual acuity at 12 months | 12 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lesya Shuba, MD PhD, Principal Investigator — CDHA Halifax Nova Scotia Canada
Locations (1):
- CDHA, Halifax, Nova Scotia, Canada